CLINICAL TRIAL: NCT06198829
Title: The Evaluation of the Relationship Between Clinical Parameters and Kinesiophobia in Patients With Femoroacetabular Impingement Syndrome
Brief Title: Evaluation of the Clinical Parameters and Kinesiophobia in Femoroacetabular Impingement Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Yagmur Kucuk, Research Assistant, Istanbul Medipol University Hospital
Other Study IDs: ACU-FTR-YK-01
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-02

CONDITIONS: Femoro Acetabular Impingement
Keywords: Pain; Kinesiophobia; Weight-Bearing; Femoracetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement; Pain; Kinesiophobia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clinical parameter assessment group: Various assessments will be conducted on patients with femoroacetabular cam impingement.
  Interventions: Other: Physical examination tests and surveys

INTERVENTIONS:
Other: Physical examination tests and surveys — Patients'hip joint range of motion range of motion, pain levels, pressure-pain threshold levels, kinesiophobia levels, and hip dysfunction levels will be measured, and the alpha angle will be evaluated on hip radiographs.

SUMMARY:
Due to the limited number of studies investigating the relationship between kinesiophobia, radiographic parameters, and clinical outcomes in patients with Femoroacetabular Impingement Syndrome (FAIS) in the literature, the aim of this study is to evaluate the relationship between kinesiophobia and clinical parameters in patients with FAIS.

DETAILED DESCRIPTION:
Femoroacetabular Impingement Syndrome (FAIS) is defined as a condition in which abnormalities in the femoral and acetabular anatomy lead to abnormal contact and mechanical forces along the joint, resulting in labral and chondral pathologies.

Symptomatic patients with Femoroacetabular Impingement Syndrome (FAIS) typically present with pain, primarily in the groin but also potentially in the lower back, hip, and posterior thigh. In addition to pain, patients may complain of a mechanically perceptible 'click' sound, locking sensation, or instability in the hip. Symptoms particularly worsen with activities such as squatting, hip rotation, sitting, climbing stairs, and prolonged sitting. The resulting symptoms lead to a decrease in functional capacities related to physical activities.

The radiographic measurements of the FAIS-Cam deformity are typically done using the alpha angle. An angle of 58 degrees or higher is considered abnormal. However, abnormal morphology is not always indicative of a pathological lesion. A holistic approach, including patient symptoms and a physical examination, is necessary for a comprehensive assessment.

In patients with Femoroacetabular Impingement Syndrome (FAIS), hip biomechanics notably change during activities such as walking, squatting, and climbing stairs. Due to pain, individuals with FAIS may exhibit protective behaviors, such as keeping the hip in flexion or adopting a Trendelenburg gait to avoid loading forces on the extremity. This situation can lead to kinesiophobia, defined as an exaggerated fear of movement and avoidance behavior based on the belief that movement may lead to injury. In patients with FAIS, it is believed that high levels of kinesiophobia are associated with lower physical function.

The participants' sociodemographic information will be recorded using a Sociodemographic Information Form. For pain assessment, the Visual Analog Scale and Algometer will be employed. Joint range of motion will be measured using the Clinometer mobile application, hip asymmetry will be assessed through the Weight Bearing Asymmetry Test using a scale, movement fear will be gauged using the Tampa Kinesiophobia Scale, and hip dysfunction will be evaluated using the Harris Hip Score. Additionally, the "Sit-to-Stand Test" will be utilized for functional measurement. The alpha angle for patients will be evaluated through pelvic anteroposterior radiography.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65
* Being diagnosed with 'cam' type femoroacetabular impingement syndrome
* Having no surgical history in the hip area and its vicinity within the last 1 year
* Having filled out the informed consent form

Exclusion Criteria:

* Having a history of psychological and mental illness
* Having another illness with symptoms that may overlap with FAI symptoms
* Refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study will include 23 patients diagnosed with FAI between the ages of 18 and 65 who have agreed to participate in the study. All participants will receive detailed information about the study, and a written informed consent form will be provided for them to voluntarily sign, indicating their acceptance of participating in the study.
  Participants will be individuals who are not candidates for surgery during the treatment process and will be selected from patients who have not undergone surgery before. The inclusion criteria involve receiving a diagnosis of 'cam' type femoroacetabular impingement syndrome through radiographic and physical examination assessments.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | One day (The assessments will be conducted once)
  The scale is a questionnaire consisting of 17 questions applicable to musculoskeletal disorders, encompassing parameters related to work-associated activities, injury/reinjury, and fear-avoidance. The scale employs a 4-point Likert rating, where 1= Strongly Disagree and 4= Strongly Agree. After reversing the scoring of items 4, 8, 12, and 16, a total score is derived. The scale yields a total score ranging from 17 to 68. A high score on the scale indicates a high level of kinesiophobia.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | One day (The assessments will be conducted once)
  The Visual Analog Scale (VAS) will be used for subjective measurement. The scale is created with a 10 cm line, with 'No Pain' written at one end and 'Unbearable Pain' at the other. The patient is asked to mark their pain intensity on this line. The portion from the 0 point to where the patient marks provides the score
Pressure-pain Threshold Levels | One day (The assessments will be conducted once)
  For objective pain measurement, an Algometer (Baseline®) will be utilized. The Algometer is a calibrated pressure device with a 1 cm round plastic-tipped end, measured in kg/cm2. It is used to measure pain associated with pressure thresholds.While applying pressure to the body with this plastic disc, the indicator needle progresses clockwise in kg. The measurement concludes when the participant feels pain, and the maximum tolerance point, obtainable in kg, is recorded.
Harris Hip Score | One day (The assessments will be conducted once)
  Harris Hip Score has been developed to measure disability in various hip problems. The questionnaire includes parameters that assess pain, function, absence of deformity, and joint range of motion. The pain domain queries the area of pain, pain intensity, activities affected by pain, and the need for medication. The function domain assesses daily activities and walking. The deformity domain includes hip movements and measurements of limb length. The joint range of motion evaluates hip mobility. The questionnaire consists of 10 items and is scored out of a maximum of 100. A higher score indicates less dysfunction.
30 Second Sit to Stand Test | One day (The assessments will be conducted once)
  The Sit-to-Stand test is employed for various purposes, including the measurement of postural control, fall risk, lower extremity strength, balance, and disability. It is suggested that the Sit-to-Stand test may serve as an indicator of lower extremity strength. The test requires a chair with a height of approximately 44 cm and back support, along with a stopwatch. When seated, the patient's feet should touch the ground, and their hands are placed crossed on their shoulders. Two practice trials are allowed before the test. The patient is instructed to stand up and sit down as quickly as possible. When standing, the hips and knees should be in full extension, and when sitting, the hips should make full contact with the chair. The number of times the patient can transition from sitting to an erect position within 30 seconds is recorded.Sitting and standing less than 10 times in 30 seconds indicates lower extremity weakness.

OTHER OUTCOMES:
Weight-Bearing Asymmetry | One day (The assessments will be conducted once)
  Two scales will be used for the assessment. Each participant's total body weight in kilograms will be recorded by having them step onto one of the scales. The scales will be used sequentially and alternately for each participant. After learning the weight of the participants, they will be placed 2 meters away from the wall with a 10 cm gap between their feet, and they will be asked to look straight ahead with one foot on each scale in an erect position. Three trials will be conducted, and the participants will be taken off the scale between trials. The average of the three measurements for each scale will be calculated, and the percentage of weight-bearing asymmetry will be determined using the following formula :
  Weight-Bearing Asymmetry Percentage = [(Load on the unaffected foot - Load on the affected foot) / Total body weight] × 100
Range of Motion | One day (The assessments will be conducted once)
  The patient's hip joint range of motion will be measured using a mobile application (Clinometer, plaincode app development and tech blog, Stephanskirchen, Germany). Wheyte et al. found that the application has excellent reliability in assessing hip extension and rotation values. The measurement will be repeated three times, and the average will be considered. For hip extension, the patient will progress from a seated position to the Modified Thomas Test position, while for internal and external rotation, the measurement will be taken with the patient in a seated position, legs hanging at 90 degrees flexion, and fixed above the knee. Measurements will be taken from the neutral position towards the direction of rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Aras Bayram, Assist.Prof., Study Director — Istanbul Medipol University School of Health Science
Locations (1):
- Acibadem Atasehir Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No